CLINICAL TRIAL: NCT04735172
Title: Exploration of Differences in Metabolite Concentrations by 7Teslas NMR Spectroscopy in Striatum and Subthalamic Nuclei in de Novo Parkinsonian Patients and Control Subjects
Acronym: METABO-NGC-7T
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AOI 2020 DURIF (METABO-NGC-7T); 2020-A03237-32 (Other: 2020-A03237-32)
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Parkinson's Disease
Keywords: De novo Parkinson's disease,; 1H Magnetic Resonance Spectroscopy,; 7 Teslas,; putamen,; Subthalamic nucleus,; glutamate,; glutamine
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- de novo PD patients (Experimental): Patients will be included:
  * suffering from idiopathic Parkinson's disease according to UKPDSBB criteria (Gibb & Lees, 1988; Hughes et al., 1992),
  * the stage of the disease is I-II according to the Hoehn and Yahr scale,
  * which do not receive dopaminergic treatment,
  * duration of disease development: 5 years,
  * without major cognitive impairment (Moca > 24)
  * men or women aged 18 to 75,
  * having understood and signed the informed consent form,
  * members of a social security scheme.
  Interventions: Other: specific MRI Acquisition (NMR spectroscopy) at 7T
- control subjects (Experimental): * subjects male or female aged 18 -75 years
  * subjects affiliated to a social security scheme.
  * volunteers who have given their written consent. They will be matched to de novo PD patients according to age, sex and level of education.
  Interventions: Other: specific MRI Acquisition (NMR spectroscopy) at 7T

INTERVENTIONS:
Other: specific MRI Acquisition (NMR spectroscopy) at 7T — The MRI protocol will be performed at 7T on a Siemens NMR imaging system (Magnetom Terra, Siemens Healthcare, Erlangen, Germany), the radio frequency emission and signal reception will be done through a head quadrature resonator (64-channel phase-array coil). To avoid motion-related artifacts, the patient will be seated in a supine position, with the arms along the body and the head immobilized using a suitable head restraint. The MR protocol will take place in two phases:
  * Acquisition of 3D multi-slice T1 and T2-weighted morphological images to identify areas of interest;
  * Acquisition of 1D RMN spectra in the right and left putamen and STN. Spectra will be acquired in volumes of interest of 15mmx15mmx15mm using a localized spectroscopy sequence with and without suppression of the water signal. Main parameters are: TR (repetition time)=3000ms; TE (echo time)=20 ms; number of repetitions=128; scan time 6min).

SUMMARY:
Initially, the exploration of brain metabolism by Nuclear Magnetic Resonance Spectroscopy (MRS) of the high magnetic field proton (1H) (11.7T) applied to acute and chronic animal models of Parkinson's disease (PD) showed glutamatergic hyperactivity within the striatum, one of the components of the basal ganglia. Interestingly, acute administration of L-dopa and acute, subchronic and chronic deep brain stimulation of the subthalamic nucleus (STN) normalizes these neurochemical profiles. Investigators also show an increase in glutamate levels in the STN ipsilateral to the substantia nigra pars compacta (SNpc) damaged by the neurotoxin, expected phenomenon, but also and surprisingly in the STN controlateral to the lesion. A degeneration of dopaminergic neurons is also observed in the controlateral SNpc at the lesion suggesting that the hyperglutamatergy of the controlateral STN to the lesion could promote neuronal death in the SNpc and thus participate in the progression and lateralization of the PD.

Using 3T MRS in PD patients, as in other studies in humans, investigators do not see changes in glutamate and glutamine levels in the putamen of Parkinsonian patients. This difference between animal and human studies can be explained:

1. by the different rate of progression between PD in humans and animal models with plasticity phenomena limiting glutamatergic hyperactivity,
2. by the effect of treatment in PD masking changes in glutamate metabolism,
3. by limiting sensitivity in the detection of metabolites (Glutamate, glutamine, GABA) at 3T.

The 7T 1H MRS improves the dispersion of chemical shifts of the metabolites studied, increases the sensitivity of the measurement, makes it possible to select regions of interest of smaller volumes (1 cm3) and thus limits the magnetic susceptibility effects that degrade the quality of the measured signal. This makes it possible to reliably separate glutamate and glutamine peaks.

In this context, investigators propose to study the metabolic changes in a homogeneous group of de novo Parkinsonian patients, naive to any treatment intended to replace the missing dopamine. The gain in spatial resolution, contrast and signal will allow better characterization of localized anomalies in small-volume structures such as basal ganglia, putamen and STN.

DETAILED DESCRIPTION:
The project presented is an open and controlled exploratory prospective study, assessing metabolic concentrations in putamen and NST left and right of treatment-naïve de novo Parkinsonian patients compared to healthy subjects. Patients will be included consecutively following the screening. Since this study is cross-sectional, a single visit will be made. De novo PD patients will be pre-selected in the departments of Neurology of the CHU of Clermont-Ferrand and Poitiers.

The inclusion visit will be carried out during a consultation during their usual follow-up in the departments of Neurology of the CHU of Clermont-Ferrand and Poitiers.

The following data will be noted: age, sex, level of study, duration of disease progression, ongoing treatments, medical history.

Patients verifying the inclusion and exclusion criteria will be definitively included and their consents will be collected.

De novo PD patients will undergo their NMR examination in the department of radiology, 7T MRI at the Poitiers hospital.

Patients will report to MRI and the following measurements will be performed:

* measurement of motor disorders by the UPDRS scale, the Hoehn and Yahr and Schwab and England score;
* acquisition of NMR images and spectra. The experimental time will be 30 minutes for the UPDRS scale and 30 minutes for the NMR exam.

Recruitment of the subjects in the control group will be carried out in the patients' family and in that of the staff of the departments of neurology and radiology.

They will be matched to de novo PD patients according to age, sex and level of education. In practice, after pre-screening the control subjects, they will be informed about the protocol, their consent will be collected. The following data will also be noted: age, sex, duration and level of study.

After verification of the inclusion and exclusion criteria, the witnesses will take the NMR examination in the Radiological Department, 7T MRI at the Poitiers University Hospital Hospital.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included:

* suffering from idiopathic Parkinson's disease according to UKPDSBB criteria (Gibb & Lees, 1988; Hughes et al., 1992),
* the stage of the disease is I-II according to the Hoehn and Yahr scale,
* which do not receive dopaminergic treatment,
* duration of disease development 5 years,
* without major cognitive impairment (Moca > 24)
* men or women aged 18 to 75,
* having understood and signed the informed consent form,
* members of a social security scheme.

Controls:

* subjects male or female aged 18 -75 years
* subjects affiliated to a social security scheme.
* volunteers who have given their written consent.

Exclusion Criteria:

Patients will be excluded:

* having a severe tremor (> 3 for a trembling sub-item of UPDRS 3) making the MR examination impossible,
* patients with "contra-indications" to an MRI exam (without administration of a gadolinium chelate): presence of metal parts in the body (electronic devices such as a pacemaker, a neurostimulator, a cochlear implant, prostheses, etc.), claustrophobia,
* taking any treatment that may interact with brain concentrations of neurotransmitters, such as all psychotropic drugs and in particular antidepressants, neuroleptics, benzodiazepines, antiepileptics,
* pregnant women,
* treated by deep brain neurostimulation,
* patients under guardianship or guardianship or protection of justice,
* patients who are excluded from another study.

Controls:

* persons suffering from progressive neurological and psychiatric pathology,
* persons with "contra-indications" to an MRI examination (without administration of a gadolinium chelate): presence of metal parts in the body (electronic devices such as a pacemaker, a neurostimulator, a cochlear implant, prostheses, etc.), claustrophobia,
* taking any treatment that may interact with brain concentrations of neurotransmitters, such as: all psychotropic drugs and in particular antidepressants, neuroleptics, benzodiazepines, antiepileptics,
* pregnant women,
* persons under guardianship or trusteeship or protection of justice,
* people who are excluded from another study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Glutamate concentration (mmol.L-1) measured in the putamen | day 90
  The concentration of glutamate present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software (Provencher 1993). It is a quantification algorithm for modelling the background noise inherent in NMR signals. This quantification method uses a database of NMR signals from the various brain metabolites simulated by quantum mechanics through their chemical and constant coupling movements (Govindaraju & al., 2000; Tkáč & al., 2005). The following 8 metabolites are included in the database: Creatine, Choline, Glutamate, Glutamine, Lactate, Myo-Inositol, N-acetylaspartate and Taurine.

SECONDARY OUTCOMES:
Glutamate concentration (mmol.L-1) measured in STN (right and left). | day 90
  The concentration of glutamate present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software (Provencher 1993). It is a quantification algorithm for modelling the background noise inherent in NMR signals. This quantification method uses a database of NMR signals from the various brain metabolites simulated by quantum mechanics through their chemical and constant coupling movements (Govindaraju & al., 2000; Tkáč & al., 2005). The following 8 metabolites are included in the database: Creatine, Choline, Glutamate, Glutamine, Lactate, Myo-Inositol, N-acetylaspartate and Taurine.
NMR spectroscopy measurements of choline,in the central grey nuclei, striatum (right and left), and NST (right and left)(mmol.L-1). | day 90
  The concentration of choline present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software
NMR spectroscopy measurements of myoinositol in the central grey nuclei, striatum (right and left), and NST (right and left)(mmol.L-1). | day 90
  The concentration of myoinositol present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software
NMR spectroscopy measurements of N-acetylaspartate in the central grey nuclei, striatum (right and left), and NST (right and left)(mmol.L-1). | day 90
  The concentration of N-acetylaspartate present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software
NMR spectroscopy measurements of creatine in the central grey nuclei, striatum (right and left), and NST (right and left)(mmol.L-1). | day 90
  The concentration of creatine present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software
NMR spectroscopy measurements of glutamine in the central grey nuclei, striatum (right and left), and NST (right and left)(mmol.L-1). | day 90
  TThe concentration of glutamine present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software
NMR spectroscopy measurements of lactate in the central grey nuclei, striatum (right and left), and NST (right and left)(mmol.L-1). | day 90
  The concentration of lactate present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software
NMR spectroscopy measurements of taurine in the central grey nuclei, striatum (right and left), and NST (right and left)(mmol.L-1). | day 90
  The concentration of taurine present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software
NMR GABA in the central grey nuclei, striatum (right and left), and NST (right and left)(mmol.L-1). | day 90
  The concentration of GABA present on the 1H NMR spectra obtained in vivo will be quantified using Lcmodel software
Severity of clinical conditions (UPDRS score) | day 90
  Clinical rating scales for PD = UPDRS

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rachel MARQUES, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Chu Clermont Ferrand, Clermont-Ferrand
  - CHU Poitiers, Poitiers